CLINICAL TRIAL: NCT03257631
Title: A PHASE 2 CLINICAL STUDY OF POMALIDOMIDE (CC-4047) MONOTHERAPY FOR CHILDREN AND YOUNG ADULTS WITH RECURRENT OR PROGRESSIVE PRIMARY BRAIN TUMORS
Brief Title: A Study of Pomalidomide Monotherapy for Children and Young Adults With Recurrent or Progressive Primary Brain Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-4047-BRN-001; U1111-1199-3348 (Registry Identifier: WHO); 2016-002903-25 (EudraCT Number)
Expanded Access: NCT03723096 (No longer available)
Record Dates: First submitted 2017-08-18; First posted 2017-08-22 (Actual); Results first posted 2019-12-10 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Central Nervous System Neoplasms; Medulloblastoma
Keywords: Pediatric; Brain Tumor; Central Nervous System Neoplasms; Glioma; High-grade glioma; HGG; Ependymoma; Medulloblastoma; DIPG; Diffuse intrinsic pontine gliomaProgressive; RecurrentPomalidomide; PomalystImnovid; CC-4047; Children
MeSH Terms: conditions — Central Nervous System Neoplasms; Medulloblastoma; Brain Neoplasms; Glioma; Ependymoma | interventions — pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pomalidomide (Experimental): Pomalidomide will administered at a starting dose of 2.6 m2/day. Pomalidomide will be provided as either a capsule (0.5 mg, 1 mg, 2 mg, 3 mg or 4 mg) or as an oral suspension (2 mg/mL).
  Interventions: Drug: Pomalidomide

INTERVENTIONS:
Drug: Pomalidomide — : Subjects will be administered pomalidomide on Days 1 to 21, followed by a 7-day rest period, of each 28-day treatment cycle and will continue treatment for up to 24 cycles or until disease progression, withdrawal of consent/assent or unresolved toxicities as described in the protocol.
  Other Names: CC-4047
Drug: Pomalidomide — Pomalidomide will be provided as gelatin capsules and as an oral suspension. The starting dose will be 2.6 mg/m²/day, administered on Days 1 to 21, followed by a 7-day rest period, of each 28-day treatment cycle.
  Other Names: CC-4047; Pomalyst®

SUMMARY:
This study will assess the efficacy, safety and tolerability of pomalidomide in children and young adults aged 1 to < 21 years with recurrent or progressive primary brain tumors in one of four primary brain tumor types: high-grade glioma (HGG), medulloblastoma, ependymoma and diffuse intrinsic pontine glioma (DIPG).

DETAILED DESCRIPTION:
The study will consist of 4 parallel groups of participants, one for each of the following primary brain tumor types: high-grade glioma, medulloblastoma, ependymoma and DIPG. A Simon's Optimal two-stage study design will be applied to each group and enrollment will occur as follows:

* Stage 1: Nine participants will be enrolled in each brain tumor type group
* Stage 2: If during Stage 1, ≥ 2 participants achieves either an objective response (either complete response or partial response) within the first 6 cycles of treatment (or within the first 3 cycles for DIPG participants), or a long-term stable disease, an additional 11 participants shall be enrolled; otherwise no additional participants will be enrolled into that group.
* If a total of 5 or more participants across all 20 participants in a given group (Stage 1 and 2) evaluable for the primary endpoint are observed as having either an objective response (either complete response or partial response) within the first 6 cycles of treatment (or within the first 3 cycles for DIPG participants) or a long-term stable disease, pomalidomide will be considered effective in that disease indication.

Once treatment has been discontinued, participants will be followed up for up to 5 years from enrollment of the last participant.

Participants who withdraw from either stage for reasons other than disease progression prior to completing Cycle 1 of study treatment will be replaced.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 1 to < 21 years of age at the time of signing the Informed Consent Form/Informed Assent Form (ICF/IAF).
2. Subject (when applicable, parental/legal representative) must understand and voluntarily sign an ICF/IAF prior to any study-related assessments/procedures being conducted.
3. Subject has received at least one prior standard therapy (or generally accepted upfront therapy if no standard exists) and have no known curative therapy.
4. Subject has a diagnosis of high-grade glioma, medulloblastoma, ependymoma or diffuse intrinsic pontine glioma (DIPG) that is recurrent or progressive. Subjects with neurofibromatosis type 1 (NF-1) associated tumors are eligible if they meet all other eligibility criteria.
5. Subject has histological verification of tumor either at the time of diagnosis or recurrence. Subjects with DIPG are exempt from histologic verification if they have typical magnetic resonance imaging (MRI) findings of DIPG
6. Subject has measurable disease defined as a tumor that is measurable in 2 perpendicular diameters on MRI. For a lesion to be considered measurable, it must be at least twice the slice thickness on MRI (ie, visible on 2 or more axial slices)
7. To document the degree of tumor at study baseline, the following scan(s) must be obtained:

   * A brain MRI with and without contrast (ie, gadolinium) and a spine MRI with contrast within 21 days prior to first dose of study treatment. For subjects on steroids, baseline MRI scans must be performed while on stable or decreasing dose of steroids for at least 5 days.
8. Subject has Karnofsky (age ≥ 16 years) or Lansky (age < 16 years) performance status score ≥ 50 at screening
9. Subject has adequate bone marrow function defined as:

   * Peripheral absolute neutrophil count (ANC) ≥ 1000/mm³
   * Platelet count ≥ 100,000/mm³ (transfusion independent defined as no platelet transfusion within 7 days and recovery from nadir)
   * Hemoglobin ≥ 8 g/dL (red blood cell [RBC] transfusion is allowed)
10. Subject has adequate renal function defined as:

    * Serum creatinine based on age/gender calculated using the Schwartz formula, or a 24-hour creatinine clearance or radioisotope glomerular filtration rate (GFR) (radioisotope or iothalamate) ≥ 70 mL/min/1.73 m².
11. Subject has adequate liver function defined as:

    * Total bilirubin ≤ 1.5 X upper limit of normal (ULN) for current age (≤ 3 X ULN if increase in bilirubin is attributable to Gilbert's Syndrome)
    * Alanine aminotransferase (ALT) (SPGT) is ≤ 3 X ULN for age
    * Serum albumin ≥ 3 g/dL
12. Subject has adequate pulmonary function defined as:

    * No evidence of dyspnea at rest
    * A pulse oximetry ≥ 93%
13. Subject has recovered from clinically significant acute treatment related toxicities from all prior therapies. Recovery is defined as a toxicity Grade ≤ 2 (common terminology criteria for adverse events [CTCAE] v. 4.03).
14. Subject has no significant worsening in clinical status for a minimum of 7 days prior to first dose of study drug.
15. Subject (and when applicable, with parental/legal representative) is willing and able to adhere to the study visit schedule and other protocol requirements.
16. Females of Childbearing Potential (FCBP) and male subjects who have reached puberty (and when applicable, with parental/legal representative) must agree to undergo physician-approved reproductive education and discuss the side effects of the study therapy on reproduction.
17. Females of childbearing potential must agree and meet the following conditions below:

    * Medically supervised (ie, performed in a clinic) pregnancy testing, including those who commit to true abstinence. Two pregnancy tests must be conducted prior to starting pomalidomide. The first pregnancy test must be performed 10 to 14 days prior to the start of pomalidomide and the second pregnancy test must be performed within 24 hours prior to starting pomalidomide. Females of childbearing potential with regular or no menstrual cycles must also agree to have pregnancy tests weekly for the first 28 days study participation, every 28 days while on study, at study treatment discontinuation, and at Day 28 following pomalidomide discontinuation. If menstrual cycles are irregular, the pregnancy testing must occur weekly for the first 28 days of study participation and then every 14 days while on study, at study treatment discontinuation visit, and at Days 14 and 28 following pomalidomide discontinuation.
    * Female subjects must, as appropriate to age and at the discretion of the study Investigator, either commit to true abstinence from heterosexual contact and/or agree to the use of two reliable forms of approved and effective contraceptive methods simultaneously. The two methods of reliable contraception must include one highly effective method (ie, oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; vasectomized partner) and one additional effective barrier method (ie, male condom, diaphragm, cervical cap) 28 days prior to starting pomalidomide, throughout the entire duration of study treatment including dose interruptions and 28 days after discontinuation of pomalidomide.
    * All male and female subjects must follow all requirements defined in the pomalidomide Pregnancy Prevention Program.
18. Male subjects must, as appropriate to age and the discretion of the study physician:

    * Practice true abstinence or agree to use a condom during sexual contact with a pregnant female or a female of child bearing potential while participating in the study, during dose interruptions and for at least 28 days following pomalidomide discontinuation, even if he has undergone a successful vasectomy or practices complete abstinence.

Exclusion Criteria:

1. Subject has a history of non-central line related thrombosis (arterial or venous), more than one prior central-line related thrombosis or known coagulopathy.
2. Subject has first degree family member with a known hereditary coagulopathy.
3. Subject is actively on anticoagulation therapy.
4. Subject has had major (per Investigator discretion) surgery, with the exception of tumor resection, within 21 days from first dose of study drug.
5. Subject has previously received (presence of any of the following will exclude a subject from enrollment):

   * Any prior treatment with pomalidomide. Subjects who have prior treatment with other immunomodulatory compounds (thalidomide, lenalidomide) are eligible if they meet all other eligibility criteria and did not have allergic reactions or other "significant toxicity" per Investigator discretion associated with lenalidomide or thalidomide use.
   * Myelosuppressive chemotherapy, immunotherapy, or any investigational agent: ≤ 21 days (≤ 42 days if a nitrosourea) prior to screening.
   * Biological (anti-neoplastic) therapy: ≤ 7 days prior to screening.
   * Immunomodulatory therapy: ≤ 28 days prior to screening.
   * Monoclonal antibody treatment and agents with known prolonged half-lives: < 3 halflives have elapsed or ≤ 28 days prior to screening, whichever is longer.
   * Prior radiation:

     * Cranial irradiation, total body irradiation (TBI), or ≥ 50% radiation of pelvis ≤ 3 months prior to screening.
     * Focal irradiation: ≤ 3 weeks prior to screening if radiation field involved a nontarget lesion; ≤ 6 weeks prior to screening if radiation field involved a target lesion.

   Note: True disease progression following prior irradiation therapy must be confirmed by Investigator prior to screening.
   * Bone marrow transplant:

     * Presence of graft versus host disease (GVHD).
     * < 6 months since allogeneic bone marrow transplant prior to screening.
     * < 3 months since autologous bone marrow/stem cell transplant prior to screening.
     * < 3 months since stem cell transplant (SCT) or Rescue without TBI with no evidence of GVHD prior to screening.
   * Radioisotopes: fluorothymidine (18FLT) ≤ 72 hours prior to first dose of study drug
6. Subject has received therapy with a known moderate to potent CYP1A2 inhibitor within 14 days or 5 half-lives of first dose of study treatment (whichever is longer).
7. Subject has received colony-stimulating growth factor(s) within 7 days prior to screening (or within 14 days if subject received polyethylene glycol formulations).
8. Subject is pregnant, breast-feeding or lactating.
9. Subject has an untreated or uncontrolled infection defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy and/or other treatment.
10. Subject has active infectious hepatitis, type A, B, or C, or chronic carriers of hepatitis C.
11. Subject has any prior history of malignancies, other than high-grade glioma, medulloblastoma, ependymoma or DIPG (Note: radiation-associated gliomas are excluded from enrollment)
12. Subject who, in the opinion of the Investigator, has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
13. Subject has any condition including the presence of laboratory abnormalities which, in the opinion of the Investigator, places the subject at unacceptable risk if he/she were to participate in the study.
14. Subject has any condition that confounds the ability to interpret data from the study.
15. Subject has symptomatic cardiac disorders (CTCAE v. 4.03 Grade 3 and 4).

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (22):
- United States (6):
  - Stanford University Cancer Center, Stanford, California
  - University Of Florida, Gainesville, Florida
  - Ann and Robert H Lurie Childrens Hospital of Chicago, Chicago, Illinois
  - Local Institution - 506, Bethesda, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Texas Children's Hospital, Houston, Texas
- France (7):
  - Local Institution - 104, Lille, Nord
  - Local Institution - 102, Lyon
  - Local Institution - 103, Marseille
  - Local Institution - 100, Paris
  - Local Institution - 106, Toulouse
  - Local Institution - 105, Vandœuvre-lès-Nancy
  - Local Institution - 101, Villejuif
- Italy (3):
  - Local Institution - 201, Genova
  - Local Institution - 200, Milan
  - Local Institution - 202, Roma
- Spain (3):
  - Local Institution - 302, Barcelona
  - Local Institution - 300, Madrid
  - Local Institution - 301, Valencia
- United Kingdom (3):
  - Local Institution - 400, Leeds
  - Local Institution - 403, London
  - Local Institution - 401, Sutton-Surrey

REFERENCES:
- [Derived] Fangusaro J, Cefalo MG, Garre ML, Marshall LV, Massimino M, Benettaib B, Biserna N, Poon J, Quan J, Conlin E, Lewandowski J, Simcock M, Jeste N, Hargrave DR, Doz F, Warren KE. Phase 2 Study of Pomalidomide (CC-4047) Monotherapy for Children and Young Adults With Recurrent or Progressive Primary Brain Tumors. Front Oncol. 2021 Jun 8;11:660892. doi: 10.3389/fonc.2021.660892. eCollection 2021. PMID 34168987
- [Derived] Fangusaro J, Mitchell DA, Kocak M, Robinson GW, Baxter PA, Hwang EI, Huang J, Onar-Thomas A, Dunkel IJ, Fouladi M, Warren KE. Phase 1 study of pomalidomide in children with recurrent, refractory, and progressive central nervous system tumors: A Pediatric Brain Tumor Consortium trial. Pediatr Blood Cancer. 2021 Feb;68(2):e28756. doi: 10.1002/pbc.28756. Epub 2020 Oct 7. PMID 33025730
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of 4 groups, for each of the following primary brain tumor types: diffuse intrinsic pontine glioma (DIPG), ependymoma, high-grade glioma, and medulloblastoma.
Pre-assignment Details: In stage 1 approximately 9 participants were to be enrolled in parallel to each group. If two or more participants in a group achieved an objective response or long-term stable disease within the first 6 cycles of treatment (within the first 3 cycles for DIPG) an additional 11 participants were to be enrolled in that group.
Groups:
- Diffuse Intrinsic Pontine Glioma; Ependymoma; High-grade Glioma; Medulloblastoma: Participants received 2.6 mg/m²/day oral pomalidomide on days 1 to 21 of each 28-day treatment cycle for up to 24 cycles or until disease progression, withdrawal of consent/assent, treatment became intolerable, or death, whichever occurred first.
Period: Overall Study
Arm/Group | Diffuse Intrinsic Pontine Glioma | Ependymoma | High-grade Glioma | Medulloblastoma
Started (The intent-to-treat population includes all enrolled participants, regardless of whether they received any treatment or not) | 11 | 9 | 23 | 10
Received Study Drug (The safety population included all participants who received at least 1 dose of study drug) | 11 | 9 | 22 | 10
Completed | 0 | 0 | 1 | 0
Not Completed | 11 | 9 | 22 | 10
Not completed — Death | 1 | 0 | 1 | 1
Not completed — Progressive Disease | 10 | 9 | 17 | 8
Not completed — Withdrawal by Parent/Guardian | 0 | 0 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat population includes all enrolled participants, regardless of whether they received any treatment or not
Groups:
- Total: Total of all reporting groups
Arm/Group | Diffuse Intrinsic Pontine Glioma | Ependymoma | High-grade Glioma | Medulloblastoma | Total
Number analyzed (Participants) | 11 | 9 | 23 | 10 | 53
Age, Continuous [Median (Full Range); unit: years] | 7.0 [4 to 12] | 12.0 [4 to 15] | 14.0 [5 to 18] | 10.0 [4 to 17] | 12.0 [4 to 18]
Age, Customized [Count of Participants; unit: Participants]
  ≥ 1 to < 6 years | 1 | 2 | 1 | 1 | 5
  ≥ 6 to < 12 years | 9 | 1 | 5 | 6 | 21
  ≥ 12 years | 1 | 6 | 17 | 3 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8 | 3 | 19
  Male | 7 | 5 | 15 | 7 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 6 | 1 | 11
  Not Hispanic or Latino | 7 | 9 | 13 | 8 | 37
  Unknown or Not Reported | 0 | 0 | 4 | 1 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 2 | 0 | 3
  Black or African American | 0 | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  White | 10 | 9 | 11 | 8 | 38
  Not Collected or Reported | 0 | 0 | 5 | 2 | 7
  Other | 0 | 0 | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Objective Response and Long-term Stable Disease
Description: The percentage of participants who achieved either an objective response, defined as a complete response (CR) or partial response (PR) in the first 6 cycles of treatment (or within 3 cycles for DIPG), or long-term stable disease (SD) defined as SD maintained for ≥ 6 cycles (≥ 3 cycles for DIPG), measured from first dose date. CR: Disappearance of all lesions and no new lesions. PR: A reduction of ≥ 50% in the size of measurable lesions, and/or persistence of non-target lesions with no progression or decrease in size. SD: A decrease of < 50% or an increase of < 25% in the size of measurable lesions and no evidence of new lesions, response does not meet the criteria for CR, PR, or progressive disease, and/or the persistence of non-target lesions with no progression or decrease in size. Progressive Disease (PD): ≥ 25% increase in the size of the measurable lesions, or the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: 6 months (first 6 cycles) or 3 months (first 3 cycles) for participants in the DIPG group
Population: The response population consisted of all enrolled participants receiving at least one cycle of pomalidomide if therapy was not discontinued earlier due to progressive disease (PD)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Diffuse Intrinsic Pontine Glioma | Ependymoma | High-grade Glioma | Medulloblastoma
Number analyzed (Participants) | 9 | 9 | 19 | 9
percentage of participants | 0 [0.0 to 33.6] | 11.1 [0.3 to 48.2] | 10.5 [1.3 to 33.1] | 0 [0.0 to 33.6]

2. Secondary Outcome: Percentage of Participants Who Achieved an Objective Response (ORR)
Description: Objective response rate was defined as the percentage of participants who achieved a complete response (CR) or partial response (PR) within the first 6 cycles of treatment (or within 3 cycles for participants in the DIPG group). Disease assessments were based on MRI and assessed by an independent central review. CR: Disappearance of all lesions and no new lesions. PR: A reduction of ≥ 50% in the size of measurable lesions compared to baseline, and/or the persistence of non-target lesions with no progression or decrease in size. Progressive Disease (PD): ≥ 25% increase in the size of the measurable lesions, or the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: 6 months (first 6 cycles) or 3 months (first 3 cycles) for participants in the DIPG group
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Diffuse Intrinsic Pontine Glioma | Ependymoma | High-grade Glioma | Medulloblastoma
Number analyzed (Participants) | 9 | 9 | 19 | 9
percentage of participants | 0 [0.0 to 33.6] | 0 [0.0 to 33.6] | 5.3 [0.1 to 26.0] | 0 [0.0 to 33.6]

3. Secondary Outcome: Percentage of Participants With Long-term Stable Disease
Description: Long-term stable disease (SD) rate was defined as the percentage of participants who achieved SD maintained for ≥ 6 cycles (or > 3 cycles for DIPG), measured from the date of first dose of treatment. Disease assessments were based on MRI and assessed by an independent central review. SD: A decrease of < 50% or an increase of < 25% in the size of measurable lesions and no evidence of new lesions, response does not meet the criteria for CR, PR, or progressive disease, and/or the persistence of non-target lesions with no progression or decrease in size. CR: Disappearance of all lesions and no new lesions. PR: A reduction of ≥ 50% in the size of measurable lesions compared to baseline, and/or the persistence of non-target lesions with no progression or decrease in size. Progressive Disease (PD): ≥ 25% increase in the size of the measurable lesions, or the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: 6 months (first 6 cycles) or 3 months (first 3 cycles) for participants in the DIPG group
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Diffuse Intrinsic Pontine Glioma | Ependymoma | High-grade Glioma | Medulloblastoma
Number analyzed (Participants) | 9 | 9 | 19 | 9
percentage of participants | 0 [0.0 to 33.6] | 11.1 [0.3 to 48.2] | 5.3 [0.1 to 26.0] | 0 [0.0 to 33.6]

4. Secondary Outcome: Duration of Response (DoR)
Description: DoR is defined as the time from the date of the first objective response (complete response [CR] or partial response [PR]) to disease progression. Participants who did not have disease progression or had not died were censored at the time of their last disease assessment or at the time of start of new anticancer therapy, whichever occurred first. Progressive disease (PD): ≥ 25% increase in the size of the measurable lesions taking as a reference the smallest disease measurement recorded since the start of protocol therapy (nadir), or the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions, or if spine MRI and/or lumbar cerebrospinal fluid (CSF) cytology were previously negative and became positive. CR: Disappearance of all lesions and no new lesions. PR: A reduction of ≥ 50% in the size of measurable lesions compared to baseline, and/or the persistence of non-target lesions with no progression or decrease in size.
Time Frame: From the first dose of pomalidomide to the date of the first documented tumor progression or death due to any cause, whichever occurs first (Up to 71 months)
Population: All enrolled participants with response (PR or CR), regardless of whether they received any treatment or not
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Diffuse Intrinsic Pontine Glioma | Ependymoma | High-grade Glioma | Medulloblastoma
Number analyzed (Participants) | 1 | 0 | 1 | 0
weeks | 12.29 [NA to NA] — 95% CI was not estimable due to insufficient number of events |  | NA [NA to NA] — Median and 95% CI were not estimable due to insufficient number of events |

5. Secondary Outcome: Kaplan-Meier Estimate of Progression-Free Survival (PFS)
Description: Progression-free survival was defined as the time from the date of first dose of pomalidomide until the date progressive disease (PD) was first observed or until the date of death due to any cause, whichever occurred first. Participants who did not have PD or had not died at the time of analysis were censored at the time of their last disease assessment or at the start of new anticancer therapy, whichever occurred first. Progressive Disease (PD): ≥ 25% increase in the size of the measurable lesions taking as a reference the smallest disease measurement recorded since the start of protocol therapy (nadir), or the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions, or if spine MRI and/or lumbar CSF cytology were previously negative and became positive.
Time Frame: as for outcome 4
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Diffuse Intrinsic Pontine Glioma | Ependymoma | High-grade Glioma | Medulloblastoma
Number analyzed (Participants) | 11 | 9 | 23 | 10
weeks | 11.43 [4.43 to 12.57] | 8.43 [5.57 to 16.14] | 7.86 [5.43 to 8.29] | 8.29 [7.29 to 18.00]

6. Secondary Outcome: Kaplan-Meier Estimate of Overall Survival (OS)
Description: Overall survival was defined as the time from the date of the first dose to the date of death (any cause). Participants who were alive were censored at the last known time that the participant was alive.
Time Frame: From the first dose of pomalidomide to the date of death due to any cause (Up to 71 months)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Diffuse Intrinsic Pontine Glioma | Ependymoma | High-grade Glioma | Medulloblastoma
Number analyzed (Participants) | 11 | 9 | 23 | 10
months | 4.86 [1.02 to 10.91] | 12.02 [2.86 to 20.90] | 5.06 [2.04 to 16.66] | 11.60 [1.74 to 35.32]

7. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Treatment-emergent adverse events were defined as any adverse events (AE) occurring from the first dose of pomalidomide until 28 days after the last dose. The severity of each AE was graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 4.03 and according to the following scale: Grade 1: Mild (transient or mild discomfort; no limitation in activity or medical intervention required); Grade 2: Moderate (mild to moderate limitation in activity, assistance may be needed; minimal medical intervention required); Grade 3: Severe (marked limitation in activity, assistance and medical intervention required, hospitalization possible); Grade 4: Life-threatening (extreme limitation in activity, significant assistance or medical intervention required, hospitalization or hospice care probable); Grade 5: Death. Drug-related AEs are those suspected by the Investigator as being related to administration of study drug.
Time Frame: From the first dose of pomalidomide until 28 days after the last dose (Up to approximately 72 months)
Population: The safety population included all participants who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Diffuse Intrinsic Pontine Glioma | Ependymoma | High-grade Glioma | Medulloblastoma
Number analyzed (Participants) | 11 | 9 | 22 | 10
Participants
  Any treatment-emergent adverse event (TEAE) | 11 | 8 | 21 | 9
  TEAE related to study drug | 5 | 7 | 14 | 8
  Serious TEAE | 9 | 4 | 14 | 4
  Serious TEAE related to study drug | 1 | 0 | 6 | 0
  Grade 3/4 TEAE | 8 | 6 | 14 | 6
  Grade 3/4 TEAE related to study drug | 3 | 2 | 10 | 4
  TEAE leading to death | 5 | 1 | 3 | 1
  TEAE leading to dose reduction | 1 | 0 | 3 | 0
  TEAE leading to dose interruption | 4 | 3 | 5 | 2
  TEAE leading to study drug discontinuation | 2 | 1 | 2 | 0

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their first dose until their study completion (up to approximately 72 months). SAEs and other AEs were assessed from first dose until 28 days after last dose (up to approximately 72 months).
Description: The number at Risk for All-cause mortality represents all enrolled participants, regardless of whether the participant received study treatment or not. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants who received at least 1 dose of pomalidomide.
Arm/Group | Diffuse Intrinsic Pontine Glioma | Ependymoma | High-grade Glioma | Medulloblastoma
All-Cause Mortality (participants affected / at risk) | 11/11 | 6/9 | 15/23 | 9/10
Serious Adverse Events (participants affected / at risk) | 9/11 | 4/9 | 14/22 | 4/10
Other Adverse Events (participants affected / at risk) | 11/11 | 8/9 | 20/22 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diffuse Intrinsic Pontine Glioma (N=11) | Ependymoma (N=9) | High-grade Glioma (N=22) | Medulloblastoma (N=10)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 2 | 1 | 2 | 1
Malaise (General disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0
Anorectal infection (Infections and infestations) | 0 | 0 | 1 | 0
Encephalitis (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Mastoiditis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 0
Respiratory syncytial virus bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 1 | 0
Dysmetria (Nervous system disorders) | 1 | 0 | 0 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 2 | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 3 | 0
Hydrocephalus (Nervous system disorders) | 0 | 2 | 2 | 0
Intracranial pressure increased (Nervous system disorders) | 1 | 0 | 1 | 0
Monoplegia (Nervous system disorders) | 0 | 0 | 0 | 1
Neurological decompensation (Nervous system disorders) | 1 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 2 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Diffuse Intrinsic Pontine Glioma (N=11) | Ependymoma (N=9) | High-grade Glioma (N=22) | Medulloblastoma (N=10)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 7 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 6 | 8 | 3
Lymphopenia (Blood and lymphatic system disorders) | 1 | 6 | 6 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 7 | 9 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3 | 8 | 3
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Blindness (Eye disorders) | 0 | 0 | 0 | 1
Conjunctival hyperaemia (Eye disorders) | 1 | 0 | 0 | 0
Mydriasis (Eye disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 1 | 5 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 5 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1 | 4 | 1
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 4 | 5 | 4
Asthenia (General disorders) | 0 | 0 | 3 | 1
Fatigue (General disorders) | 2 | 1 | 4 | 2
Gait disturbance (General disorders) | 0 | 1 | 0 | 1
General physical health deterioration (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 2 | 0
Pyrexia (General disorders) | 2 | 1 | 2 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0
Eye infection (Infections and infestations) | 1 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 1 | 0 | 0
Molluscum contagiosum (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 1
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 0
Parotitis (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 1 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 3 | 1 | 0
Rhinovirus infection (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 4 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 3 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 2 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 1 | 0
Ataxia (Nervous system disorders) | 2 | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 3 | 0
Headache (Nervous system disorders) | 3 | 4 | 5 | 3
Hemiparesis (Nervous system disorders) | 0 | 0 | 2 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1 | 1 | 0
Muscle spasticity (Nervous system disorders) | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 1
Pyramidal tract syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1
VIth nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Personality change (Psychiatric disorders) | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Tonsillar inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 3 | 2 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Pallor (Vascular disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2017-12-20): https://cdn.clinicaltrials.gov/large-docs/31/NCT03257631/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-20): https://cdn.clinicaltrials.gov/large-docs/31/NCT03257631/SAP_001.pdf